CLINICAL TRIAL: NCT04171557
Title: Bicycling and Mortality Among Individuals With Diabetes in the European Prospective Investigation Into Cancer and Nutrition (EPIC)
Brief Title: Bicycling and Mortality Among Individuals With diabetesNutrition (EPIC)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Mathias Ried-Larsen, Senior Researcher, Rigshospitalet, Denmark
Other Study IDs: Bicycling and Diabetes (17-25)
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Diabete Mellitus
Keywords: Exercise; Physical Activity; Bicycling
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes at the baseline assessement in EPIC: Self-reported and confirmed diabetes (validated by a second source (at least 1), including repeated self-report, contact with physician, linkage to register later point, intake of diabetes medicine, registration of diabetic chiropody, baseline glycated hemoglobin>=6.0%, five annual blood glucose measurements or two blood glucose measurements per year for five consecutive years) cases were included in the analyses. No information is available to distinguish between type 1 and type 2 diabetes across the population but type 1 is rare by comparison.
  Interventions: Behavioral: Bicycling

INTERVENTIONS:
Behavioral: Bicycling — Total bicycling is reported in categories of: (0 - reference), (>0 to <60), (≤60 to >150), (≤150 to < 300) and (≥300) minutes/week

SUMMARY:
The primary aim of the study is to study the relationship between overall bicycling and all-cause mortality and secondarily cardiovascular disease mortality among individuals with diabetes from European countries. A secondary aim will be to study the relation of change in bicycling to all-cause mortality and cardiovascular disease mortality.

DETAILED DESCRIPTION:
AIMS The primary aim of the study is to study the relationship between overall bicycling and all-cause mortality and secondarily cardiovascular disease mortality among individuals with diabetes from European countries. A secondary aim will be to study the relation of change in bicycling to all-cause mortality and cardiovascular disease mortality.

METHODS Study design and setting The study is a nested cohort study in European Prospective Investigation into Cancer and Nutrition (EPIC) cohort. In EPIC, 29 centers in 10 western European countries have collected information on nutrition, lifestyle, anthropometrics and medical history from more than 521 000 study individuals participating in this prospective cohort study. Dietary, medical history and lifestyle were assessed by questionnaires. Blood samples from the participants were taken at the study centers. Baseline (first examination) information was collected 1992-2000 and second examination for exposure has since been obtained at least once in every cohort. Exposure data has subsequently, to the two examinations, been linked to information on vital status and on cause of death were obtained through record linkages with national, regional or local registers, regional health departments, physicians or hospitals, active follow-up or health insurance.

Study population This nested prospective cohort study, sampled individuals with prevalent diabetes in the EPIC cohorts at the baseline assessments in the years 1992-2000. Self-reported and confirmed diabetes (validated by a second source (at least 1), including repeated self-report, contact with physician, linkage to register later point, intake of diabetes medicine, registration of diabetic chiropody, baseline glycated hemoglobin>=6.0%, five annual blood glucose measurements or two blood glucose measurements per year for five consecutive years) cases were included in the analyses. No information is available to distinguish between type 1 and type 2 diabetes across the population but type 1 is rare by comparison. The nested cohort for this study comprised 12,848 individuals with self-reported and/or confirmed diabetes. Mean (SD) follow-up time was 14.6 (4.8) years. Among the 12,848 prevalent diabetes cases, 5,809 cases were confirmed at baseline as described above.

For further detail, please see the predefined statistical analysis plan (SAP). It can be accessed through the url: http://aktivsundhed.dk/images/docs/SAPMRL.pdf

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or self-reported diabetes at first examination

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See Statistical Analysis Plan
Sampling Method: Non-Probability Sample
Enrollment: 12848 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
All-cause Mortality | From 0 years and up to 17 years or until death from any cause, whichever comes first.
  0 (Alive at follow-up) or 1 (Death at follow-up)

SECONDARY OUTCOMES:
Cause specific mortality: Cardiovascular | From 0 years and up to 17 years or until death from any cause, whichever comes first.
  0 (Alive at follow-up) or 1 (Death at follow-up: cause being International Classification of Diseases, Injuries, and Causes of Death, Tenth Revision, I00-I99 )

OTHER OUTCOMES:
Cause specific mortality: Cardiovascular | From 4-6 years (second examination) after 0 years (first examination) and up to 12 years or until death from any cause, whichever comes first.
  0 (Alive at follow-up) or 1 (Death at follow-up: cause being International Classification of Diseases, Injuries, and Causes of Death, Tenth Revision, I00-I99 )
All-cause Mortality | From 4-6 years (second examination) after 0 years (first examination) and up to 12 years or until death from any cause, whichever comes first.
  0 (Alive at follow-up) or 1 (Death at follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, PhD, Principal Investigator — Copenhagen University Hospital, Centre for Physical Activity Research
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Request for individual patient data should be directed to the International Agency for Research on Cancer (IARC)
  The predefined statistical analyses plan is available (see link)